CLINICAL TRIAL: NCT03597659
Title: PheWAS of a Polygenic Predictor of Thyroid Function
Acronym: PHETHYR
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-18-09
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Thyroid; Genetic Predisposition to Disease
MeSH Terms: conditions — Thyroid Diseases; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BioVU-Emerge EHR cohort: A primary EHR population derived from the eMERGE Phase I & II Network (n=16,924), a consortium of medical centers using EHRs as a tool for genomic research, and from Vanderbilt University Medical Center's (VUMC) BioVU resource (n=20,230).
  BioVU is VUMC's de-identified collection of patients whose DNA was extracted from discarded blood and linked to phenotypes through a de-identified EHR.
  All subjects were born prior to 1990 and fell within 4 standard deviations for each of the first 2 principal components based on common single nucleotide variants (SNVs) for the subset of subjects self-identified as "White, non-Hispanic".
  Interventions: Genetic: phenome-wide association study (PheWAS)

INTERVENTIONS:
Genetic: phenome-wide association study (PheWAS) — Phenome-wide association study (PheWAS) identifying clinical diagnoses associated with a polygenic predictor of TSH levels identified by a previously published genome-wide association study (GWAS) which included North American and European participants. A phenome-wide scanning of 1,318 phenotypes will be performed, using a cohort of 37,154 North American individuals of European ancestry with electronic-health-record (EHR) data.

SUMMARY:
Performing a phenome-wide association study (PheWAS) identifying clinical diagnoses associated with a polygenic predictor of Thyroid stimulating hormone (TSH) levels identified by a previously published genome-wide association study (GWAS). PheWAS will be applied in an electronic-health-record (EHR) cohort including North American (n: 37,154) and European participants using 1,318 phenotypes.

DETAILED DESCRIPTION:
Applying a genetic predictor of thyroid stimulating hormone levels to an electronic-health-record cohort to verify associations with thyroid disorders as positive controls, and identify new associations .

ELIGIBILITY:
Inclusion Criteria:

* Being part of the eMERGE Phase I & II Network
* Being part of the BioVU resource
* Falling within 4 standard deviations for each of the first 2 principal components based on common single nucleotide variants (SNVs) for the subset of subjects self-identified as "White, non-Hispanic"

Exclusion Criteria:

* born after 1990

Ages: 28 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A primary electronic health record population derived from the eMERGE Phase I & II Network (n=16,924), and from Vanderbilt University Medical Center's (VUMC) BioVU resource (n=20,230). All subjects born prior to 1990 and falling within 4 standard deviations for each of the first 2 principal components based on common single nucleotide variants (SNVs) for the subset of subjects self-identified as "White, non-Hispanic".
  Thyroid Stimulating Hormone(TSH)-Population subgroup: Subjects of European Ancestry in BioVU who did not have any ICD-9 or ICD-10 codes for thyroid diseases and who had thyroid stimulating hormone (TSH) measurements that fell within the clinically normal reference range.
Sampling Method: Non-Probability Sample
Enrollment: 37154 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
thyroid disorders associated with a polygenic predictor of thyroid stimulating hormone levels | population inclued in the eMERGE Phase I & II Network or BioVU resource until 1 july 2018
  All relevants statisticals associations between a defined polygenic predictor of TSH and thyroids disorders

SECONDARY OUTCOMES:
Clinical diagnoses associated with a polygenic predictor of TSH levels | population inclued in the eMERGE Phase I & II Network or BioVU resource until 1 july 2018
  All relevants statisticals associations between a defined polygenic predictor of thyroid stimulating hormone and clinical diagnoses

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salem JE, Shoemaker MB, Bastarache L, Shaffer CM, Glazer AM, Kroncke B, Wells QS, Shi M, Straub P, Jarvik GP, Larson EB, Velez Edwards DR, Edwards TL, Davis LK, Hakonarson H, Weng C, Fasel D, Knollmann BC, Wang TJ, Denny JC, Ellinor PT, Roden DM, Mosley JD. Association of Thyroid Function Genetic Predictors With Atrial Fibrillation: A Phenome-Wide Association Study and Inverse-Variance Weighted Average Meta-analysis. JAMA Cardiol. 2019 Feb 1;4(2):136-143. doi: 10.1001/jamacardio.2018.4615. PMID 30673079